CLINICAL TRIAL: NCT06799923
Title: Possibilities of Use Magnetic Resonance Imaging (MRI)-Guided Laser Interstitial Thermal Therapy (LITT) in Treatment of Medically Intractable Tremor
Brief Title: Possibilities of Use MRI-Guided Laser Interstitial Thermal Therapy in Medically Intractable Tremor
Acronym: PossibiLITT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Rouen (Other); University Hospital, Caen (Other); Central Hospital Saint Quentin (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2021_843_0110
Record Dates: First submitted 2024-09-24; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-09

CONDITIONS: Laser Interstitial Thermal Therapy; Parkinson Disease; Essential Tremor; Movement Disorders; MRI
Keywords: laser interstitial thermal therapy; Parkinson Disease; Essential Tremor; Movement Disorders; MRI
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parkinson's disease (Experimental): Patients 18 years age or older with Parkinson's disease or essential tremor and tremor resistant to medical therapy with a contraindication to deep brain stimulation or refusal deep brain stimulation
  Interventions: Procedure: laser electrode

INTERVENTIONS:
Procedure: laser electrode — A laser electrode is implanted surgically in the ventral and inteermediary nucleus of the thalamus (VIM).

SUMMARY:
Medically intractable tremors are a common difﬁcult clinical situation. Deep brain stimulation decreases Parkinson's disease tremor and essential tremor, but not all patients are candidates from a diagnostic, medical, or social standpoint, prompting the need for alternative surgical strategies. Less invasive lesional brain surgery (thalamotomy) procedures by radio-surgery or MRI-guided focused ultrasound have emerged and have proven to be effective in these third-line indications. Recently, a new technology has emerged allowing the performance of minimally invasive lesion surgeries by MRI-Guided Laser Interstitial Thermal Therapy (MRIg-LITT). MRIg-LITT has been shown to be effective and safe in management of epilepsies and brain tumors. However, no study has evaluated MRIg-LITT for performing thalamotomy in medically intractable tremor.In a pilot study, the investigators propose to evaluate the effect and safety of unilateral thalamotomy by MRIg-LITT in the management of medically intractable tremor of parkinsonian or essential origin.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years age or older with Parkinson's disease or essential tremor and tremor resistant to medical therapy with a contraindication to deep brain stimulation or refusal deep brain stimulation

Exclusion Criteria:

* Contraindication to MRI
* Contraindication to general anesthesia
* Patient unable to give their free and informed consent because of cognitive or psychiatric disorders
* Brain anatomical abnormalities not allowing intervention
* Adults protected (guardianship, curators) or deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Variation of total body weight from baseline | at 72 hours
  To assess the impact of UF prescription guided by the ECW/TBWat ratio on weight loss, a comparison of TBW (∆TBW) between the two groups will be conducted. The ∆TBW is the difference between the initial TBW at H0 and the TBW at H72.

SECONDARY OUTCOMES:
cumulative fluid balance | at 72 hours
  Cumulative fluid balance is the difference between fluids administered (intravenous fluids, blood products, enteral nutrition, replacement fluid from RRT) and fluid loss (weight loss from RRT, urine output, blood loss, enteral loss, and losses through drains). It is calculated using the cumulative net UF from RRT and the hospital software (DianeRéa, Bowmedical, version 4.8.11.22887) over the period from H0 to H72.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Salouël, France

IPD SHARING:
Plan to Share IPD: No